CLINICAL TRIAL: NCT03404193
Title: A Phase II Study of Venetoclax in Combination With 10-Day Decitabine in Newly Diagnosed Elderly or Relapsed/Refractory Acute Myeloid Leukemia and Relapsed High-Risk Myelodysplastic Syndrome and Blastic Plasmacytoid Dendritic Cell Neoplasm
Brief Title: Venetoclax and Decitabine in Treating Participants With Relapsed/Refractory Acute Myeloid Leukemia or Relapsed High-Risk Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0912; NCI-2018-00752 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0912 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Blastic Plasmacytoid Dendritic Cell Neoplasm; Chronic Myelomonocytic Leukemia; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndrome; Recurrent Acute Biphenotypic Leukemia; Recurrent Acute Myeloid Leukemia; Recurrent Blastic Plasmacytoid Dendritic Cell Neoplasm; Recurrent Chronic Myelomonocytic Leukemia; Recurrent Mixed Phenotype Acute Leukemia; Refractory Acute Myeloid Leukemia; Refractory Blastic Plasmacytoid Dendritic Cell Neoplasm; Refractory Chronic Myelomonocytic Leukemia; Refractory Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Blastic Plasmacytoid Dendritic Cell Neoplasm; Leukemia, Myelomonocytic, Chronic; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes | interventions — Decitabine; Injections; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, venetoclax) (Experimental): Participants receive decitabine IV over 1 hour on days 1-10 and may also receive decitabine on days 1-5 after achieving complete remission/complete remission with incomplete count recovery during consolidation/maintenance. Participants also receive venetoclax PO daily on days 1-28 of cycle 1 and on days 1-21 of subsequent cycles. Treatment repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Decitabine; Other: Laboratory Biomarker Analysis; Drug: Venetoclax

INTERVENTIONS:
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase II trial studies how well venetoclax and decitabine work in treating participants with acute myeloid leukemia that has come back or does not respond to treatment, or with high-risk myelodysplastic syndrome that has come back. Drugs used in chemotherapy, such as venetoclax and decitabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the overall response rate (ORR) of venetoclax in combination with 10-day decitabine in patients with refractory/relapsed acute myeloid leukemia (AML); elderly (> 60 year old) patients with newly diagnosed AML not eligible for intensive chemotherapy; patients with high-risk myelodysplastic syndrome (MDS) with bone marrow blasts between 10% and 20%, relapsed or refractory to prior hypomethylating agent (HMA) therapy, or chronic myelomonocytic leukemia (CMML) with bone marrow blasts >= 10% regardless of prior therapy; AML patients with prior history of MDS or CMML who received therapy for the MDS or CMML and progressed to AML, and younger patients with newly diagnosed AML with poor risk complex karyotype and/or TP53 deletions/mutations and patients with blastic plasmacytoid dentritic cell neoplasm (BPDCN).

SECONDARY OBJECTIVES:

I. To determine the duration of response, disease-free survival (DFS), and overall survival (OS) of patients with refractory/relapsed AML treated with this combination.

II. To determine the number of patients who achieve a hematologic improvement (HI) in platelets, hemoglobin, or absolute neutrophil count (ANC) and the number of patients who achieve > 50% reduction in blasts on therapy with venetoclax/10-day decitabine.

III. To determine the safety of venetoclax in combination with 10-day decitabine in patients with refractory/relapsed AML.

IV. To determine the number of patients who transition towards stem cell transplantation upon achieving response with the combination venetoclax/10-day decitabine regimen.

V. To determine the incidence of infectious complications per cycle with venetoclax in combination with 10-day decitabine.

EXPLORATORY OBJECTIVES:

I. To investigate possible relationships between baseline protein and gene expression signatures/mutation profile and BH3 profiling in predicting clinical response to the combination.

II. To characterize the pharmacokinetic (PK) profiles of venetoclax in combination with decitabine and antifungals in plasma samples.

OUTLINE:

Participants receive decitabine intravenously (IV) over 1 hour on days 1-10 and may also receive decitabine on days 1-5 after achieving complete remission/complete remission with incomplete count recovery during consolidation/maintenance. Participants also receive venetoclax orally (PO) daily on days 1-28 of cycle 1 and on days 1-21 of subsequent cycles. Treatment repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up every 3 to 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with AML, BPDCN, biphenotypic or bilineage leukemia (including a myeloid component) or mixed phenotype acute leukemia (MPAL) who have failed prior therapy; patients with AML should have failed prior therapy or have relapsed after prior therapy; patients with isolated extramedullary AML are eligible
* Elderly (> 60 year old) patients with newly diagnosed AML, BPDCN, or mixed phenotype acute leukemia (MPAL) not eligible for intensive chemotherapy
* Patients with newly diagnosed AML with poor risk complex karyotype and/or TP53 deletions/mutations equal or younger than 60 year old
* AML or BPDCN patients with prior history of MDS or CMML who received any therapy or no therapy for the MDS or CMML and progressed to AML, are eligible at the time of diagnosis of AML regardless of any prior therapy for MDS; the World Health Organization (WHO) classification will be used for AML
* Patients with high-risk MDS with bone marrow blasts between 10% and 20%, relapsed or refractory to prior hypomethylating agent (HMA) therapy, defined as prior receipt of 4 cycles of HMA therapy with failure to attain a response, or relapse after prior response to HMA therapy; patients with high risk chronic myelomonocytic leukemia (CMML) with bone marrow blasts >= 10% regardless of prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 3
* White blood cell count =< 10,000
* Adequate renal function including creatinine < 2 unless related to the disease
* Adequate hepatic function including total bilirubin < 2 x upper limit of normal (ULN) unless increase is due to Gilbert's disease or leukemic involvement
* Alanine aminotransferase (ALT) < 3 x ULN unless considered due to leukemic involvement
* Provision of written informed consent
* Oral hydroxyurea and/or one dose of cytarabine (up to 2 g/m^2) for patients with rapidly proliferative disease is allowed before the start of study therapy and while the patient is on active study treatment through cycle 1, as needed, for clinical benefit and after discussion with the principal investigator (PI); concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted
* Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment
* Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment; males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment

Exclusion Criteria:

* Patients having received any prior BCL2 inhibitor therapy
* Patients with t(15;17) karyotypic abnormality or acute promyelocytic leukemia (French-American-British [FAB] class M3-AML)
* Patients with symptomatic CNS leukemia or patients with poorly controlled CNS leukemia
* Active and uncontrolled comorbidities including active uncontrolled infection, uncontrolled hypertension despite adequate medical therapy, active and uncontrolled congestive heart failure New York Heart Association (NYHA) class III/IV, clinically significant and uncontrolled arrhythmia as judged by the treating physician
* Patients with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C
* Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | Up to 4 cycles (112 days)
  Will be defined as the proportion of patients who had CR (complete remission), CRp (complete remission with incomplete platelet recovery), CRi (complete remission with incomplete count recovery), PR (partial response) or marrow clearance of blasts within 3 months of treatment initiation among adult patients with acute myeloid leukemia (AML); and complete remission (CR), partial remission (PR) or marrow CR (mCR) lasting at least 4 weeks for patients with myelodysplastic syndrome (MDS). Descriptive statistics including plots, mean, median and standard deviations will be used to summarize data. Will estimate the ORR for the combination treatment, along with the 95% confidence interval. The association between ORR and patient's clinical characteristics will be examined by Wilcoxon's rank sum test or Fisher's exact test, as appropriate.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 5 years
  Toxicity type, severity and attribution will be summarized for each patient using frequency tables.
Duration of response | Up to 5 years
  Will be estimated using the method of Kaplan-Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log rank tests.
Disease free survival | Up to 5 years
  Will be estimated using the method of Kaplan-Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log rank tests.
Overall survival | Up to 5 years
  Will be estimated using the method of Kaplan-Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log rank tests.

OTHER OUTCOMES:
Biomarker analysis | Baseline
  Baseline protein, gene expression signatures/mutation profile and BH3 profiling will be summarized with descriptive statistics. The correlation with endpoints of anti tumor activity will be explored where possible.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Venugopal S, Maiti A, DiNardo CD, Qiao W, Ning J, Loghavi S, Daver NG, Kadia TM, Rausch CR, Alvarado Y, Ohanian M, Sasaki K, Short NJ, Takahashi K, Yilmaz M, Ravandi F, Kantarjian HM, Konopleva MY. Prognostic impact of conventional cytogenetics in acute myeloid leukemia treated with venetoclax and decitabine. Leuk Lymphoma. 2021 Dec;62(14):3501-3505. doi: 10.1080/10428194.2021.1973675. Epub 2021 Sep 3. No abstract available. PMID 34474640
- [Derived] Kim K, Maiti A, Loghavi S, Pourebrahim R, Kadia TM, Rausch CR, Furudate K, Daver NG, Alvarado Y, Ohanian M, Sasaki K, Short NJ, Takahashi K, Yilmaz M, Tang G, Ravandi F, Kantarjian HM, DiNardo CD, Konopleva MY. Outcomes of TP53-mutant acute myeloid leukemia with decitabine and venetoclax. Cancer. 2021 Oct 15;127(20):3772-3781. doi: 10.1002/cncr.33689. Epub 2021 Jul 13. PMID 34255353
- [Derived] Maiti A, DiNardo CD, Wang SA, Jorgensen J, Kadia TM, Daver NG, Short NJ, Yilmaz M, Pemmaraju N, Borthakur G, Bose P, Issa GC, Ferrajoli A, Jabbour EJ, Jain N, Garcia-Manero G, Ohanian M, Takahashi K, Montalban-Bravo G, Masarova L, Burger JA, Thompson PA, Verstovsek S, Sasaki K, Andreeff M, Rausch CR, Montalbano KS, Pierce S, Qiao W, Ning J, Kantarjian HM, Konopleva MY, Ravandi F. Prognostic value of measurable residual disease after venetoclax and decitabine in acute myeloid leukemia. Blood Adv. 2021 Apr 13;5(7):1876-1883. doi: 10.1182/bloodadvances.2020003717. PMID 33792630
- [Derived] Venugopal S, Maiti A, DiNardo CD, Loghavi S, Daver NG, Kadia TM, Rausch CR, Alvarado Y, Ohanian M, Sasaki K, Short NJ, Takahashi K, Yilmaz M, Ravandi F, Kantarjian HM, Konopleva MY. Decitabine and venetoclax for IDH1/2-mutated acute myeloid leukemia. Am J Hematol. 2021 May 1;96(5):E154-E157. doi: 10.1002/ajh.26122. Epub 2021 Feb 19. No abstract available. PMID 33580980
- [Derived] Laribi K, Baugier de Materre A, Sobh M, Cerroni L, Valentini CG, Aoki T, Suzuki R, Takeuchi K, Frankel AE, Cota C, Ghez D, Le Calloch R, Pagano L, Petrella T. Blastic plasmacytoid dendritic cell neoplasms: results of an international survey on 398 adult patients. Blood Adv. 2020 Oct 13;4(19):4838-4848. doi: 10.1182/bloodadvances.2020002474. PMID 33027528
- [Derived] DiNardo CD, Maiti A, Rausch CR, Pemmaraju N, Naqvi K, Daver NG, Kadia TM, Borthakur G, Ohanian M, Alvarado Y, Issa GC, Montalban-Bravo G, Short NJ, Yilmaz M, Bose P, Jabbour EJ, Takahashi K, Burger JA, Garcia-Manero G, Jain N, Kornblau SM, Thompson PA, Estrov Z, Masarova L, Sasaki K, Verstovsek S, Ferrajoli A, Weirda WG, Wang SA, Konoplev S, Chen Z, Pierce SA, Ning J, Qiao W, Ravandi F, Andreeff M, Welch JS, Kantarjian HM, Konopleva MY. 10-day decitabine with venetoclax for newly diagnosed intensive chemotherapy ineligible, and relapsed or refractory acute myeloid leukaemia: a single-centre, phase 2 trial. Lancet Haematol. 2020 Oct;7(10):e724-e736. doi: 10.1016/S2352-3026(20)30210-6. Epub 2020 Sep 5. PMID 32896301
- See also: MD Anderson Cancer Center — http://www.mdanderson.org